CLINICAL TRIAL: NCT03130166
Title: Intracorporeal Versus Extracorporeal Anastomosis in Robotic Right Colectomy - a Double-blinded Randomized Controlled Trial
Brief Title: INtracorporeal Versus EXtracorporeal Anastomosis in Robotic Right Colectomy
Acronym: INEXA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Niclas Dohrn, MD., Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCT0001
Record Dates: First submitted 2017-04-23; First posted 2017-04-26 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Colonic Cancer
Keywords: Postoperative pain; Postoperative recovery; Intracorporeal anastomosis; Robotic right colectomy
MeSH Terms: conditions — Colonic Neoplasms; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracorporeal anastomosis (Experimental): Patients undergo robotic right colectomy with intracorporeal anastomosis.
  Interventions: Procedure: Intracorporeal anastomosis
- Extracorporeal anastomosis (Active Comparator): Patients undergo robotic right colectomy with extracorporeal anastomosis.
  Interventions: Procedure: Extracorporeal anastomosis

INTERVENTIONS:
Procedure: Intracorporeal anastomosis — Use of intracorporeal anastomosis technique
  Arms: Intracorporeal anastomosis
Procedure: Extracorporeal anastomosis — Use of the conventional extracorporeal anastomosis technique
  Arms: Extracorporeal anastomosis

SUMMARY:
Right-sided colonic cancer is treated with right-sided colectomy, predominantly performed as minimally invasive surgery with extracorporeal anastomosis (ECA). In recent years a new technique with intracorporeal anastomosis (ICA) has emerged and it is thought that ICA is less invasive and thereby has the potential to improve the postoperative course of right colonic cancer patients.

The objective of this study is to compare robotic right colectomy with either ICA or ECA in a randomized controlled setting.

ELIGIBILITY:
Inclusion Criteria:

All patients scheduled for robotic right colectomy due to colonic cancer are eligible for inclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
Postoperative recovery | 1 month
  Questionnaire of Recovery 15 (QoR-15)

SECONDARY OUTCOMES:
Time fo first flatus | 1 month
Time to first bowel movement | 1 month
Length of hospital stay | 1 month
Morbidity | 1 month
Mortality | 1 month
Postoperative pain | 1 month
Heart Rate Variability | 2 days
  Continuously ECG-monitoring intraoperatively and postoperatively
"Timed up and go"-test | 2 days
Ortostatic hypotension test | 2 days
Spirometry and PEF - test | 2 days
  Postoperative pulmonary function
Postoperative opioid usage | 1 month
Whole blood gene expression profiling | 1 month
  Measuring changes in expression of ROS and immulogical genes due to surgery.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Herlev Hospital, Herlev, Copenhagen
  - Sealand University Hospital, Roskilde

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dohrn N, Oppermann C, Yikilmaz H, Laursen M, Khesrawi F, Clausen FB, Jakobsen HL, Brisling S, Lykke J, Eriksen JR, Klein MF, Gogenur I. The effect of intracorporeal versus extracorporeal anastomosis in robotic right colectomy on perianastomotic perfusion: a substudy to a multicenter RCT. Langenbecks Arch Surg. 2022 Dec;407(8):3577-3586. doi: 10.1007/s00423-022-02693-4. Epub 2022 Sep 28. PMID 36171282
- [Derived] Dohrn N, Yikilmaz H, Laursen M, Khesrawi F, Clausen FB, Sorensen F, Jakobsen HL, Brisling S, Lykke J, Eriksen JR, Klein MF, Gogenur I. Intracorporeal Versus Extracorporeal Anastomosis in Robotic Right Colectomy: A Multicenter, Triple-blind, Randomized Clinical Trial. Ann Surg. 2022 Nov 1;276(5):e294-e301. doi: 10.1097/SLA.0000000000005254. Epub 2021 Oct 13. PMID 35129520
- [Derived] Dohrn N, Klein MF, Gogenur I. Intracorporeal versus extracorporeal anastomosis in right colectomy - a protocol for a randomised trial. Dan Med J. 2021 Apr 20;68(5):A09200710. PMID 33913415